CLINICAL TRIAL: NCT02771717
Title: Does a Low Exhaled Nitric Oxide Level Exclude a Clinical Benefit From Inhaled Corticosteroids in Suspected Asthma: A Randomised, Placebo Controlled Trial
Brief Title: Low Exhaled NO and ICS in Suspected Asthma
Acronym: LowNO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16013
Record Dates: First submitted 2016-04-28; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Pulmicort) (Experimental): Low dose inhaled corticosteroid.
  Interventions: Drug: Budesonide (Pulmicort)
- Placebo - dummy inhaler (Placebo Comparator): Placebo - dummy inhaler
  Interventions: Drug: Placebo - dummy inhaler

INTERVENTIONS:
Drug: Budesonide (Pulmicort) — Budesonide (Pulmicort) - inhaled low dose inhaled steroid - I puff to be taken twice daily
  Arms: Budesonide (Pulmicort)
Drug: Placebo - dummy inhaler — Placebo - dummy inhaler to be taken 1 puff twice daily.
  Other Names: Placebo
  Arms: Placebo - dummy inhaler

SUMMARY:
The purpose of this study is to determine whether a low exhaled nitric oxide reading (<27ppb) is a good predictor of a negative response to inhaled steroid treatment for patients with symptoms suggestive of asthma.

DETAILED DESCRIPTION:
At the first visit, which will take place at either at the GP surgery or the Nottingham Respiratory Research Unit (NRRU) informed written consent for the study will be obtained. The patients will then have an exhaled NO measurement, spirometry, venepuncture (for Full Blood Count and research blood - if consent obtained) taken and complete an Asthma Control Questionnaire (ACQ), Medical Research Council dyspnoea scale (MRC) and Leicester Cough Questionnaire (LCQ). All procedures will be carried out by the NRRU research nurse.

The investigators may use the NRRU existing database of research volunteers to recruit as necessary and also the respiratory clinics held at the NUH. If patients from clinics are recruited they will be initially approached by their usual care doctor and an information sheet will be sent / given to them accordingly.

If all the inclusion criteria are met and none of the exclusion criteria, the patients will be randomised to receive either a placebo inhaler, to be taken one puff twice daily, or a low dose inhaled steroid treatment, Budesonide 200mcgs via Turbuhaler one puff twice daily, for 3 months. Dr Tim Harrison will be prescribing the inhalers and they will be dispensed from the Nottingham City Hospital Clinical Trials Pharmacy and delivered/given to the patient by the research nurses.

Participants will be asked to return for follow up visits at 4 weeks, 8 weeks and 12 weeks following randomisation. At these follow up visits, exhaled NO, spirometry and the 3 questionnaires will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over.
2. Asthma suspected by GP/Practice Nurse
3. Must be able to give informed consent
4. Exhaled Nitric Oxide reading <27ppb
5. FEV1 >70% predicted

Exclusion Criteria:

1. Patients requiring oral steroid treatment on visit to GP/Practice nurse
2. Use of oral prednisolone or antibiotics within last 4 weeks
3. Already using an inhaled corticosteroid
4. Any other clinically significant co-morbidity.
5. Expectant or breast feeding mothers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Difference in Asthma Control Questionnaire (ACQ-7) between the inhaled steroid and placebo group adjusted for differences in baseline. The ACQ will measure the level of asthma control in the ICS and placebo group. | overall 12 weeks
  Data will be collect via questionnaire at each visit. A change in ACQ-7 of 0.5 is considered clinically important.

SECONDARY OUTCOMES:
Difference in FEV1 between inhaled steroid and placebo groups adjusted for differences in baseline. | overall 12 weeks
  FEV1 will be measured in Litres.
Measure cough symptoms with the LCQ between ics and placebo group adjusted for differences in baseline. | overall 12 weeks
  A minimal important difference in LCQ is 1.3. This will be assessed using this validated, self-reported measure of quality of life for cough.
Difference in a subjective measurement of MRC dyspnoea scale. | overall 12 weeks
  This is a subjective scale of breathlessness graded 1-5 (5 being most breathless). This will be assessed from baseline measurements.

OTHER OUTCOMES:
The incidence of asthma exacerbations will be recorded for each group and compared. | 12 weeks
  The number of asthma exacerbations will be captured from verbal feedback from specific patient questioning at study visits.
The deterioration in asthma control as measured by ACQ-7 and compared between groups. | 12 weeks
  deterioration in asthma control will be captured from the ACQ- 7

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dr Harrison, MD, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: No